CLINICAL TRIAL: NCT07085611
Title: Study of the Neutralizing Power of Serum Antibodies - 2 (PNAS-2)
Brief Title: Neutralizing Power of Serum Antibodies - 2
Acronym: PNAS-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUO-2024-22
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: COVID-19; SARS-CoV-2 Viraemia; Monkey Pox; Vaccination; Serum; Mucosal Immunity
Keywords: Neutralizing antibodies; SARS-CoV-2; Monkeypox; Vaccination; Serum; Mucosal immunity
MeSH Terms: conditions — COVID-19; Mpox, Monkeypox | interventions — Specimen Handling; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Each participant receives the treatment (vaccine or monoclonal antibody) indicated by clinical practice. Samples (blood ± nasal swab) are collected at maximum 13 timepoints over 60 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving vaccines and/or monoclonal antibodies (Other): Participants receive standard-of-care SARS-CoV-2 and/or MPXV vaccines or monoclonal antibodies. This study does not assign the treatment but collects biosamples to assess antibody response.
  Interventions: Other: Sample collection (blood and optional nasal swab)

INTERVENTIONS:
Other: Sample collection (blood and optional nasal swab) — Venous blood collection (2 tubes of 6 mL) and optional nasal swab at each visit. Aliquots analyzed for neutralizing activity against SARS-CoV-2 and MPXV using validated assays at Institut Pasteur

SUMMARY:
Severe forms of COVID-19 and Monkeypox affect immunocompromised and comorbid individuals. Vaccination and monoclonal antibody therapies induce neutralizing antibodies. This neutralizing power is recognized as a correlate of protection against a new infection. This study aims to describe the neutralizing power of serum and nasal antibodies over time, in relation to SARS-CoV-2 and MPXV vaccines or treatments received.

DETAILED DESCRIPTION:
This is a monocentric, longitudinal, descriptive study aiming to measure and describe the evolution of the humoral immune response (serum and nasal) to SARS-CoV-2 and MPXV, following any vaccination or administration of monoclonal antibodies. Samples are collected over a maximum 60-month period per participant to assess the durability of neutralizing activity.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Patients receiving or scheduled to receive anti-SARS-CoV-2 and/or anti-MPXV vaccines or monoclonal antibodies
* Patients have provided written informed consent

Exclusion Criteria:

* Persons under guardianship or curatorship
* Persons under legal protection,
* Persons persons deprived of liberty
* Persons not affiliated to a social security scheme
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2030-08-22 (Estimated); Study Completion 2035-07-11 (Estimated)

PRIMARY OUTCOMES:
Serum neutralizing antibody evolution (anti-SARS-CoV-2 and anti-MPXV) over time | Up to 60 months
  S-Fuse and S-Flow tests performed on collected serum samples at each visit

SECONDARY OUTCOMES:
Mucosal (nasal) neutralizing antibody response and MPXV serology over time | Up to 60 months
  Nasal antibody neutralization (anti-MPX) and serum MPXV neutralization assessed using validated Pasteur Institute protocols
Mucosal (nasal) neutralizing antibody response and SARS-CoV-2 serology over time | Up to 60 months
  Nasal antibody neutralization (anti-SARS-CoV-2) and serum SARS-CoV-2 neutralization assessed using validated Pasteur Institute protocols

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PRAZUCK, Dr, Principal Investigator — CHU Orléans
Locations (1):
- CHU Orléans, Orléans, France

REFERENCES:
- [Background] Grzelak L, Temmam S, Planchais C, Demeret C, Tondeur L, Huon C, Guivel-Benhassine F, Staropoli I, Chazal M, Dufloo J, Planas D, Buchrieser J, Rajah MM, Robinot R, Porrot F, Albert M, Chen KY, Crescenzo-Chaigne B, Donati F, Anna F, Souque P, Gransagne M, Bellalou J, Nowakowski M, Backovic M, Bouadma L, Le Fevre L, Le Hingrat Q, Descamps D, Pourbaix A, Laouenan C, Ghosn J, Yazdanpanah Y, Besombes C, Jolly N, Pellerin-Fernandes S, Cheny O, Ungeheuer MN, Mellon G, Morel P, Rolland S, Rey FA, Behillil S, Enouf V, Lemaitre A, Creach MA, Petres S, Escriou N, Charneau P, Fontanet A, Hoen B, Bruel T, Eloit M, Mouquet H, Schwartz O, van der Werf S. A comparison of four serological assays for detecting anti-SARS-CoV-2 antibodies in human serum samples from different populations. Sci Transl Med. 2020 Sep 2;12(559):eabc3103. doi: 10.1126/scitranslmed.abc3103. Epub 2020 Aug 17. PMID 32817357
- [Background] Planas D, Bruel T, Grzelak L, Guivel-Benhassine F, Staropoli I, Porrot F, Planchais C, Buchrieser J, Rajah MM, Bishop E, Albert M, Donati F, Prot M, Behillil S, Enouf V, Maquart M, Smati-Lafarge M, Varon E, Schortgen F, Yahyaoui L, Gonzalez M, De Seze J, Pere H, Veyer D, Seve A, Simon-Loriere E, Fafi-Kremer S, Stefic K, Mouquet H, Hocqueloux L, van der Werf S, Prazuck T, Schwartz O. Sensitivity of infectious SARS-CoV-2 B.1.1.7 and B.1.351 variants to neutralizing antibodies. Nat Med. 2021 May;27(5):917-924. doi: 10.1038/s41591-021-01318-5. Epub 2021 Mar 26. PMID 33772244
- [Background] Hubert M, Guivel-Benhassine F, Bruel T, Porrot F, Planas D, Vanhomwegen J, Wiedemann A, Burrel S, Marot S, Palich R, Monsel G, Diombera H, Gallien S, Lopez-Zaragoza JL, Vindrios W, Taieb F, Fernandes-Pellerin S, Delhaye M, Laude H, Arowas L, Ungeheuer MN, Hocqueloux L, Pourcher V, Prazuck T, Marcelin AG, Lelievre JD, Batejat C, Levy Y, Manuguerra JC, Schwartz O. Complement-dependent mpox-virus-neutralizing antibodies in infected and vaccinated individuals. Cell Host Microbe. 2023 Jun 14;31(6):937-948.e4. doi: 10.1016/j.chom.2023.05.001. Epub 2023 May 5. PMID 37196656